CLINICAL TRIAL: NCT01078948
Title: A Double-blind Sham Controlled Trial of Transcranial Direct Current Stimulation (tDCS) in Treating Refractory Major Depressive Disorder (MDD)
Brief Title: Transcranial Direct Current Stimulation (tDCS) in the Treatment of Major Depressive Disorder (MDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Director, Brain Stimulation Treatment and Research Program, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 157/2007
Record Dates: First submitted 2008-02-25; First posted 2010-03-02 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Major Depressive Disorder
Keywords: tDCS; transcranial direct current stimulation; major depression; double-blind; randomized; placebo-controlled; treatment
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active 2mA tDCS (Experimental): The stimulator will be used to deliver anodal stimulation to the left prefrontal cortex and cathodal stimulation to the right prefrontal cortex. The placement of the anode is proposed to enhance activity in the left frontal cortex; the cathode aims to reduce activity in the right prefrontal cortex.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): The system setup is identical to that of active tDCS; however, the stimulator will be turned off after 30 seconds.
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Delivery of mild current to specified brain regions.
  Other Names: Stimulator CX-6650 (Rolf Schneider Electronics, Germany)

SUMMARY:
The project will investigate the use of a novel neuromodulatory technique, transcranial direct current stimulation (tDCS) in the treatment of patients with major depressive disorder.

Hypothesis 1: Active tDCS will improve depressive symptomology to a significantly greater degree than sham treatment.

Hypothesis 2: Active tDCS will be well tolerated and free of major side effects.

DETAILED DESCRIPTION:
Major depression is a disorder with major clinical and economic significance locally and internationally. It is a disorder of high prevalence and results in substantial disease burden and health-care costs. Critically, a significant percentage of patients, usually estimated at around 30%, fail to respond to standard treatments (Fitzgerald 2003). Techniques, such as repetitive transcranial magnetic stimulation (rTMS), are being investigated widely for the treatment of this disorder, with considerable success in recent years (Fitzgerald, Benitez et al. 2006; Hasey 2001). However, TMS equipment is expensive and requires specialized application. Additionally, TMS is associated with some side-effects (e.g. seizures). Given that depression occurs in all cultures and countries, there would be considerable value in developing a low-cost, non-invasive technique that can be applied in a wide variety of settings and which has already been shown to have some efficacy in MDD (Boggio et al. 2007).

The proposed study will be a randomized, double blind, placebo-controlled (i.e., sham stimulation vs. active tDCS), longitudinal, treatment outcome trial. Individuals with MDD will be randomized to 1 of 2 treatment conditions. These will be:

1. Active 2mA tDCS: in this condition, 1 stimulator will be used with anodal stimulation to the left prefrontal cortex and cathodal stimulation to the right prefrontal cortex. The placement of anodal stimulation is proposed to enhance activity in the left frontal cortex; the cathode aims to reduce activity in the right prefrontal cortex.
2. Sham treatment: the system setup is identical to that of active tDCS, but the stimulator will be turned off after 30 seconds.

A total of 15 treatments will be administered to all participants over 3 weeks (one per working day). Individuals will be randomized on a computer-generated list. Clinical raters and patients will be blind to the treatment condition. Clinical ratings well be conducted prior to and after the treatment course (i.e., after 3 weeks). All subjects randomized to sham treatment will be offered active treatment at the end of the acute treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Competent to consent
* Have a diagnosis of Major Depressive Disorder and are currently experiencing a Major Depressive Episode as confirmed by the SCID-IV
* Treatment resistant, defined as a failure to achieve a clinical response, or an inability to tolerate, at least two trials of antidepressant medication of sufficient dose for at least 6 weeks
* Aged 18 to 75.
* Concomitant medications including: benzodiazepines, mood stabilizers antidepressants and anticholinergics will be allowed. Since carbamazepine has been shown to interfere with the effects of anodal tDCS, potential participants taking it will not be suitable for inclusion in the trial.

Exclusion Criteria:

* DSM-IV history of substance abuse or dependence in the last 6 months
* A major and/or unstable medical or neurologic illness
* Currently taking carbamazepine
* Pregnancy
* History of seizures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAMD), 17-item version | Baseline and at 3 weeks
  The Hamilton Depression Scale (HAMD) is a clinician administered test measuring the severity of depressive symptoms in adults and children.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Daskalakis, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Blumberger DM, Tran LC, Fitzgerald PB, Hoy KE, Daskalakis ZJ. A randomized double-blind sham-controlled study of transcranial direct current stimulation for treatment-resistant major depression. Front Psychiatry. 2012 Aug 17;3:74. doi: 10.3389/fpsyt.2012.00074. eCollection 2012. PMID 22912618
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research